CLINICAL TRIAL: NCT04004078
Title: An Individualized Administration Research of Voriconazole Based on CYP2C19 Gene Polymorphism and Therapeutic Drug Monitoring in Chinese Patients With Invasive Pulmonary Infection
Brief Title: An Individualized Administration Research of Voriconazole Based on CYP2C19 Gene Polymorphism and TDM
Status: Completed | Type: Observational
Sponsor: People's Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, LIjuan Zhou, Principal Investigator, People's Hospital of Zhengzhou University
Other Study IDs: zhou750423
Record Dates: First submitted 2019-06-26; First posted 2019-07-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Invasive Fungal Infection
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Group A: Non-gene directed group：Voriconazole was intravenously administered 2 times at the loading dose of 6mg/Kg at 12h intervals , followed by maintenance dosing 4mg/Kg at 12h intervals . Voriconazole was oral administered 2 times at the loading dose of 400mg or 200mg（weight>40Kg or <40Kg）at 12h intervals , followed by maintenance dosing 200mg or 100mg（weight>40Kg or <40Kg）. Voriconazole was sequential therapy administered 2 times at the loading dose of 6mg/Kg at 12h intervals , followed by maintenance dosing 200mg or 100mg（weight>40Kg or <40Kg）.
  Interventions: Device: other antifungal agents,breathing machine
- Group B: Gene directed group（UMs and EMs）：The dosage of the drug was the same as that of the non-gene-directed group for patients with UMs，EMs.
  Interventions: Device: other antifungal agents,breathing machine
- Group C: Gene directed group（IMs）：The dosage of the drug was the same as that of the non-gene-directed group for patients with IMs.
  Interventions: Device: other antifungal agents,breathing machine
- Group D: Gene directed group（PMs）： Voriconazole was intravenously administered 2 times at the loading dose of 4mg/Kg at 12h intervals , followed by maintenance dosing 3mg/Kg at 12h intervals . Voriconazole was oral administered 2 times at the loading dose of 200mg or 100mg（weight>40Kg or <40Kg）at 12h intervals , followed by maintenance dosing 100mg . Voriconazole was sequential therapy administered 2 times at the loading dose of 4mg/Kg at 12h intervals , followed by maintenance dosing 100mg.
  Interventions: Device: other antifungal agents,breathing machine

INTERVENTIONS:
Device: other antifungal agents,breathing machine — If treatment failure for patients in group A，group B，group C and group D，change other antifungal agents(Amphotericin B for Injection,25mg,North China Pharmaceutical Co., Ltd or Caspofungin Acetate for lnjection,50mg and 70mg Cancidas®). Mechanical ventilation((EVITA 4, Dräger Medical Equipment (Shanghai) Co.,Ltd) was adopte.Treatment failure was defined as no improvement or worse of clinical symptoms, laboratory data, requiring change of antifungal agents therapy.

SUMMARY:
This was a prospective clinical study that all voriconazole-treated adult Chinese patients with invasive pulmonary infection admitted to Zhengzhou Central Hospital affiliated to Zhengzhou University from March 2018 to April 2020.

DETAILED DESCRIPTION:
This was a prospective clinical study that all voriconazole-treated adult Chinese patients with invasive pulmonary infection admitted to Zhengzhou Central Hospital affiliated to Zhengzhou University from March 2018 to April 2020. Patients were included who met the following criteria:(1)age≥18 years old, (2)Diagnosis of invasive fungal infection,(3)written informed consent was obtained from each patients,(4)At least one steady trough concentration blood sample was taken from each patient.

Patients were excluded who fulfilled any of the following criteria:(1) patients who are allergic to voriconazole or have poor compliance, (2) use other antifungal drugs during the use of VCZ, (3) do not qualify for blood sampling monitored by blood concentration, (4) patients with severe liver function impairment (ALT and AST before VCZ treatment are greater than 5 times the normal upper limit, TBIL is greater than 3 times the normal upper limit), 5) pregnant or lactating women, (6) with incomplete clinical data collection, (7) have participated in other clinical trials in the past three months.

Grouping: 1) The patients were grouped according to CYP2C19 gene detection, they were divided into gene-directed group and non-gene-directed group; 2) According to the effect of treatment, the patients were divided into effective group and ineffective group; 3) According to whether patients had adverse reactions, they were divided into group A (adverse reactions) and group B (no adverse reactions). The clinical indicators and detection values of each group were recorded, respectively.

Loading Dosage of administration and treatment regimen : All the selected patients were treated with VCZ. Dose of administration is shown for gene-directed group and non-gene-directed group below. The maintenance dosage was increased or decreased appropriately up to target Cmin range (0.5μg/ml~5.0μg/ml).

According to CYP2C19 gene detection, phenotypes were classified as ultrarapid metabolisers(UMs)，extensive metabolisers(EMs) ，intermediate metabolisers(IMs) and poor metabolisers(PMs).

Dose of administration and treatment regimen according to CYP2C19 gene detection:(1)Non- gene directed group：Voriconazole was intravenously administered 2 times at the loading dose of 6mg/Kg at 12h intervals , followed by maintenance dosing 4mg/Kg at 12h intervals . Voriconazole was oral administered 2 times at the loading dose of 400mg or 200mg（weight>40Kg or <40Kg）at 12h intervals , followed by maintenance dosing 200mg or 100mg（weight>40Kg or <40Kg）. Voriconazole was sequential therapy administered 2 times at the loading dose of 6mg/Kg at 12h intervals , followed by maintenance dosing 200mg or 100mg（weight>40Kg or <40Kg）. (2) Gene directed group: The dosage of the drug was the same as that of the non-gene-directed group for patients with UMs，EMs and IMs. For the patients with PMs，Voriconazole was intravenously administered 2 times at the loading dose of 4mg/Kg at 12h intervals , followed by maintenance dosing 3mg/Kg at 12h intervals . Voriconazole was oral administered 2 times at the loading dose of 200mg or 100mg（weight>40Kg or <40Kg） at 12h intervals , followed by maintenance dosing 100mg . Voriconazole was sequential therapy administered 2 times at the loading dose of 4mg/Kg at 12h intervals , followed by maintenance dosing 100mg.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years old
* Diagnosis of invasive fungal infection
* written informed consent was obtained from each patients
* At least one steady trough concentration blood sample was taken from each patient

Exclusion Criteria:

* patients who are allergic to voriconazole or have poor compliance
* use other antifungal drugs during the use of VCZ
* do not qualify for blood sampling monitored by blood concentration
* patients with severe liver function impairment (ALT and AST before VCZ treatment are greater than 5 times the normal upper limit, TBIL is greater than 3 times the normal upper limit)
* pregnant or lactating women,
* with incomplete clinical data collection
* have participated in other clinical trials in the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All voriconazole-treated adult Chinese patients with invasive pulmonary infection were admitted to Zhengzhou Central Hospital affiliated to Zhengzhou University from March 2018 to April 2020.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Serum voriconazole trough concentrations | 0.5 hour before voriconazole administration on the Thirdth or sixth day
  If all patients were administrated by loading dose, voriconazole trough samples were taken immediately 30 minutes before Voriconazole administration on the Third day. If all patients were not administrated by loading dose, voriconazole trough samples were taken immediately 30 minutes before Voriconazole administration on the sixth day. Blood samples for 2-3 mL were collected in blood-collection tubes without any additives and centrifuged at 3500 rpm for 10min. Serum trough concentrations (Cmin) were determined by a high-performance liquid chromatography method as previously described. The detections were completed in Translational Medicine Center of Zhengzhou Central Hospital affiliated to Zhengzhou University.

SECONDARY OUTCOMES:
The difference of average Cmin among group A, group B, group C and group D | From March 2018 to April 2020
  The differences were counted among group A, group B, group C and group D by measuring each person's Cmin.
The correlation between Cmin and CRP, IL-6 and PCT | From March 2018 to April 2020
  The correlation between Cmin and CRP, IL-6 and PCT by Pear's correlation analysis .CRP,IL-6 and PCT were completed before initiation ,after voriconazole therapy on day 3,7 and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
The effect of voriconazole on liver injury biomarkers | From March 2018 to April 2020
  The effects of different level of voriconazole-Cmin (<0.5,0.5-5,and>5μg/ml ) on liver injury biomarkers( ALT,AST,ALP and GGT ).The differences among 3groups were compared using one-way analysis of variance /post(Scheffe) test.They were determined before initiation ,after voriconazole therapy on day 3,7 and completion of voriconazole therapy in Zhengzhou city clinical inspection center.
Determination of Predictors of voriconazole Cmin | From March 2018 to April 2020
  The voriconazole Cmin variation may be influenced by many factors. A backward multiple linear regression model was performed for determination of predictors of voriconazole Cmin.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou Central Hospital affiliated to Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No